CLINICAL TRIAL: NCT03995355
Title: Clinical Evaluation of an Investigational Lipid Drop in Non-contact Lens Wearing Patients
Status: Completed | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6328
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Results first posted 2022-11-14 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Test Eye Drops (Experimental): Eligible subjects that are non-contact lens wearers will be randomized to the Test group throughout the duration of the study.
  Interventions: Device: 9618X investigational lipid eye drops
- Control Eye Drops (Active Comparator): Eligible subjects that are non-contact lens wearers will be randomized to the Control group throughout the duration of the study.
  Interventions: Device: Blink® Tears

INTERVENTIONS:
Device: 9618X investigational lipid eye drops — Test Eye Drops
  Arms: Test Eye Drops
Device: Blink® Tears — Control Eye Drops
  Arms: Control Eye Drops

SUMMARY:
This is a double-masked, randomized, bilateral, 2-Arm parallel group study. Subjects are scheduled for 3 study visits (screening/baseline, 7-Day and 30-Day follow-up visits) over a period of one month.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. Subjects must be at least 18 years of age and no more than 69 years of age (inclusive).
  2. Subjects must be non-contact lens wearers.
  3. Subjects must achieve visual acuity of 20/30 or better in each eye, either unaided or best corrected.
  4. Subjects must possess a functional/usable pair of spectacles and bring them to every visit (only if applicable - to the investigators discretion).
  5. Self-reported symptoms of ocular dryness or irritation and/or the use of artificial tears in the last 3 months.
  6. Subjects must read, understand, and sign the Statement of Informed Consent.
  7. Subjects must appear able and willing to adhere to the instructions set forth in this clinical protocol.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or breast-feeding.
  2. Diabetes.
  3. Any ocular or systemic allergies or disease which may interfere with the clinical trial (at the investigator's discretion).
  4. Any systemic disease, autoimmune disease, or use of medication which may interfere with the clinical trial (at the investigator's discretion).
  5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
  6. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA scale.
  7. Any active ocular abnormalities/conditions that may interfere with the clinical trial (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection, etc.).
  8. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology.
  9. History of any ocular or corneal surgery (e.g. RK, PRK, LASIK).
  10. Participation in any pharmaceutical or medical device related clinical trial within 30 days prior to study enrollment.
  11. History of binocular vision abnormality or strabismus.
  12. Habitual wearers of soft contact lenses in the past 1 month or rigid gas permeable lens within the past 3 months.
  13. Current habitual use of Prescription Medicines to treat dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator).
  14. Employees of investigational clinic (investigator, coordinator, and technician, etc.) or family member of an employee of the clinical site by self-report.

In addition to the above criteria, patients with any allergy or sensitivity to ingredients that this product may contain (Castor Oil, Polyoxyl 40 Hydrogenated Castor Oil, Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate, Purified Water) should not participate in the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Premier Vision, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Derived] Donnenfeld E, Coats J, Barbour K, Ryan R, Joshi NR, Periman LM. Efficacy and safety of a lipid-containing artificial tear compared with a non-lipid containing tear: a randomized clinical trial. BMC Ophthalmol. 2024 Oct 8;24(1):442. doi: 10.1186/s12886-024-03688-z. PMID 39379885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 161 subjects were enrolled in this study. Of those enrolled, 158 subjects were dispensed a test article while 3 subjects failed to meet all eligibility criteria. Of those dispensed, 155 subjects completed the study while 3 subjects were discontinued.
Groups:
- Test (Investigational Lipid Eye Drop): Subjects randomized to the Test eye drops throughout the entire duration of the study.
- Control (Blink Tears Eye Drops): Subjects that instilled the Control eye drops throughout the study
Period: Overall Study
Arm/Group | Test (Investigational Lipid Eye Drop) | Control (Blink Tears Eye Drops)
Started | 77 | 81
Completed | 75 | 80
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Scheduling Issues | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Investigational Lipid Eye Drop) | Control (Blink Tears Eye Drops) | Total
Number analyzed (Participants) | 77 | 81 | 158
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (14.51) | 48.8 (13.8) | 47.8 (14.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 56 | 114
  Male | 19 | 25 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 10 | 24
  White | 63 | 68 | 131
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 77 | 81 | 158

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Ocular Comfort (30-Day)
Description: Subjective overall ocular comfort was assessed at baseline, and at the 30-Day follow-up using a Visual Analogue Scale (VAS) ranging from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline ocular comfort score was calculated as 30-Day follow-up score minus Baseline score. Change from Baseline VAS Scores range from -100 to 100, where higher change from baseline comfort scores indicates better performance. The average change from baseline comfort score for each Arm was report.
Time Frame: Baseline and 30-Day Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Test (Investigational Lipid Eye Drops): Subjects that instilled the Test eye drops throughout the study.
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 63 | 67
Units on a scale | 21.4 (24.51) | 10.0 (26.01)
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Non-Inferiority — Subjective overall comfort was analyzed using linear mixed model. Statistical inference was made based on the 95% confidence interval constructed for the least square mean difference; Linear Mixed Model Analysis; Least square mean difference = 11.3, 95% CI 2-sided [2.6 to 20.1], Standard Error of Mean 4.44 — Least square mean difference was calculated as Test minus Control

2. Secondary Outcome: Change From Baseline Ocular Comfort (7-Day)
Description: Subjective overall ocular comfort was assessed at baseline, and at the 7-Day follow-up using a Visual Analogue Scale (VAS) ranging from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline ocular comfort score was calculated as 7-Day follow-up score minus Baseline score. Change from Baseline VAS Scores range from -100 to 100, where higher change from baseline comfort scores indicates better performance. The average change from baseline comfort score for each Arm was report.
Time Frame: Baseline and 7-Day Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 63 | 67
Units on a scale | 14.3 (24.02) | 11.7 (21.23)
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least square mean difference = 2.6, 95% CI 2-sided [-5.3 to 10.4], Standard Error of Mean 3.97 — Least square mean difference was calculated as Test minus Control

3. Secondary Outcome: Number of Subject Eyes That Reported Ocular Symptoms
Description: Subjects were reported whether they experienced any ocular symptoms, problems or complaints (yes/no) by eye. Ocular symptoms were assessed for each subject eye at all study visits (scheduled and unscheduled). The number of eyes that experience ocular symptoms or complaints was reported for the 7- and 30-Day follow-up.
Time Frame: 7-Day Follow-up and 30-Day Follow-up
Population: All subjects/eyes who were that administered any test article excluding subjects who dropped out prior to administering any test article.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 77 | 81
Number analyzed (Eyes) | 154 | 162
Eyes
  7-Day Follow-up | 33 | 37
  30-Day Follow-up | 21 | 21
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Other; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 0.967, 95% CI 2-sided [0.528 to 1.770] — Odds ratio was calculated as Test over Control. No difference was concluded if 1 fall within the 95% confidence interval for the odds ratio
Statistical Analysis 2: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); 30-Day follow-up; Test type: Other; Generalized linear Mixed Model Analysis; Odds Ratio (OR) = 1.160, 95% CI 2-sided [0.610 to 2.203] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Number of Subject Eyes That Experience Grade 2 or Higher Corneal Staining
Description: Corneal staining was analyzed using the FDA grading scale (ie, Grade 0 = None, Grade 1 = Trace, Grade 2 = Mild, Grade 3 = Moderate and Grade 4 = Severe). These responses were categorized into a binary outcome as 1 if any Grade 2 or higher corneal staining was observed or otherwise 0 is recorded. Subjects with multiple events were counted only once for the analysis purpose.
Time Frame: 7-Day Follow-up and 30-Day Follow-up
Population: All subjects who were administered any test article excluding subjects who dropped out prior to administering any test article.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 77 | 81
Number analyzed (Eyes) | 154 | 162
Eyes
  7-Day Follow-up | 1 | 2
  30-Day Follow-up | 2 | 0
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Other; Fisher Exact; Odds Ratio (OR) = 1.601, 95% CI 2-sided [0.178 to 19.616] — Odds ratio was calculated as Test over Control

5. Secondary Outcome: Change From Baseline Ocular Vision (7-Day)
Description: Subjective overall ocular vision was assessed at baseline, dispensing and 7-Day follow-up using a Visual Analogue Scale (VAS) from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline ocular vision score was calculated as 7-Day follow-up score minus Baseline score. Change from Baseline VAS Scores range from -100 to 100, where higher change from baseline vision scores indicates better performance. The average change from baseline vision score for each Arm was report.
Time Frame: Baseline and 7 Day-Day Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 63 | 67
Units on a scale | 13.3 (23.23) | 5.2 (19.23)
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Other; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Net) = 8.0, 95% CI 2-sided [0.7 to 15.4], Standard Error of Mean 3.73 — Least square mean difference was calculated as Test minus Control

6. Secondary Outcome: Change From Baseline Ocular Vision (30-Day)
Description: Subjective overall ocular vision was assessed at baseline, dispensing and 30 Day follow-up using a Visual Analogue Scale (VAS) from 0 (extremely uncomfortable) to 100 (extremely comfortable). The change from baseline ocular vision score was calculated as 30-Day follow-up score minus Baseline score. Change from Baseline VAS Scores range from -100 to 100, where higher change from baseline vision scores indicates better performance. The average change from baseline vision score for each Arm was report.
Time Frame: Baseline and 30 Day Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Test (Investigational Lipid Eye Drops) | Control (Blink Tears Eye Drops)
Number analyzed (Participants) | 63 | 67
Units on a scale | 14.2 (22.52) | 4.9 (21.55)
Statistical Analysis 1: Comparison: Test (Investigational Lipid Eye Drops) vs Control (Blink Tears Eye Drops); Test type: Other; Linear Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Mean Difference (Net) = 9.3, 95% CI 2-sided [1.7 to 17.0], Standard Error of Mean 3.86 — Least square mean difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throught the entire duration of the study. Approximately 30 Days per subject.
Arm/Group | Test (Investigational Lipid Eye Drop) | Control (Blink Tears Eye Drops)
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/81
Serious Adverse Events (participants affected / at risk) | 1/77 | 1/81
Other Adverse Events (participants affected / at risk) | 0/77 | 0/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Investigational Lipid Eye Drop) (N=77) | Control (Blink Tears Eye Drops) (N=81)
Corneal Edema Due to Trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pancreatitis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03995355/Prot_SAP_000.pdf